CLINICAL TRIAL: NCT02957253
Title: Effects on Liver Cirrhotic Patient's Health Related Quality of Life by a Nurse-led Clinic: A Multicenter Randomized Controlled Trial
Brief Title: Effects on Liver Cirrhotic Patients' by a Nurse-led Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Fundation of Ester Åsberg-Lindbergs memories, Falun; Sweden (Unknown); Center for Clinical Research Dalarna, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hjorth, Principal investigator, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/146
Record Dates: First submitted 2016-10-18; First posted 2016-11-07 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Liver Cirrhosis
Keywords: Quality of care; Health related quality of life; Nurse-led clinic; Health economics
MeSH Terms: conditions — Liver Cirrhosis | interventions — Risk Factors; Self Care; Nutritional Status; Practice Patterns, Nurses'

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention (CI) (Experimental): Compensated intervention (CI). Nurse-led clinic one time per year. Focus on Life style and risk factors.
  Interventions: Other: risk factors; Other: lifestyle; Other: Nurse-led clinic
- Control (CC) (No Intervention): Compensated Control (CC)
- Intervention (DI) (Experimental): Decompensated intervention (DI). Nurse-led clinic two times every month to every third month. Focus on Lifestyle, risk factors, nutrition, selfcare and psychosocial needs
  Interventions: Other: risk factors; Other: self-care; Other: nutrition; Other: lifestyle; Other: psychosocial needs; Other: Nurse-led clinic
- Control (DC) (No Intervention): Decompensated Control (DC)

INTERVENTIONS:
Other: risk factors — monitoring risk factors due to deterioration of the liver disease
  Arms: Intervention (CI); Intervention (DI)
Other: self-care — information and motivation to adherence to self-care instructions and medical treatment
  Arms: Intervention (DI)
Other: nutrition — nutritional assessment and activities to prevent malnutrition
  Arms: Intervention (DI)
Other: lifestyle — motivation of lifestyle changes essential for disease progress and
  Arms: Intervention (CI); Intervention (DI)
Other: psychosocial needs — psychosocial care.
  Arms: Intervention (DI)
Other: Nurse-led clinic — compensated disease once yearly, decompensated disease twice a month to every third month
  Arms: Intervention (CI); Intervention (DI)

SUMMARY:
This study compare the effects of traditional follow-up by physician with a combined follow-up alternately by physician and nurse-led clinic. The main variable is; health related quality of Life. Participants are randomized into control group or intervention group.

DETAILED DESCRIPTION:
The incidence of liver cirrhosis in Sweden increase mostly due to life style factors. A large need of care is common in the end stage of the disease. Nurse-led clinics for other groups of patients, e.g. coronary heart disease, have shown high quality which has resulted in an established part of the follow-up.

This study is a randomized controlled study at six Swedish hospitals to study the effect of a changed follow-up process for liver cirrhotic patients by adding a nurse-led clinic to follow up by physician. The intervention implies a larger extend of nursing interventions at the outpatient clinic to increase the patient's quality of life, quality of care and reduce the need of inpatient care.

A few hospitals in Sweden offers a nurse-led clinic for liver cirrhotic patients, the interest in other hospitals are raising. Though there is a lack of evidence in nursing intervention within this population and it is still unknown what the effects are for the individual or on the health economy.

ELIGIBILITY:
Inclusion Criteria:

* within the last 24 months diagnosed liver cirrhosis based on clinical investigation, laboratory findings, histology, magnetic resonance imaging, computer tomography, ultrasound or elastography
* followed at one of the six Gastroenterology departments

Exclusion Criteria:

* Insufficient knowledge of the Swedish language
* Persistent hepatic ecephalopathy grades 2-4
* Comorbidity: Chronic obstructive pulmonary disease grade 3-4, Coronary heart disease New York Heart Association Functional Classification class 3-4, Dementia, Actual advanced cancer, Stroke with sequelae, Severe psychiatric disease, Renal failure requiring dialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Health related quality of life | At baseline after 12 and 24 months
  Patient survey using the instrument from Research and development, RAND 36-item heath survey

SECONDARY OUTCOMES:
Clinical examination of presence of ascites | At baseline after 12 and 24 months
  Severity of ascites is grouped as none, mild or severe
Child-Pugh scale | At baseline after 12 and 24 months
  Liver cirrhosis specific calculator to measure long time survival
Presence of Hepatic encephalopathy | At baseline after 12 and 24 months
  Paper and pencil test the psychometric hepatic encephalopathy score (PHES)
Health literacy | At baseline after 12 and 24 months
  Standardized interview of a table of contents using the instrument The newest vital sign (NVS)
Model of end stage liver disease (MELD-score) | At baseline after 12 and 24 months
  A liver cirrhosis specific calculator to assess short time survival rate
Risk assessment of malnutrition using the instrument the Royal free hospital - nutritional prioritizing tool | At baseline after 12 and 24 months
  A liver cirrhosis specific instrument will be used to assess the risk of malnutrition. The risk is subdivided into low, moderate or high risk.
Changes in patients experienced Quality of care | At baseline after 12 and 24 months
  Patient survey using the instrument Quality of care from the the patient's perspective (QPP)
Health care consumption | through study completion, 24 months
  Medical Review of inpatient and outpatient care

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rönnblom, Professor, Study Chair — Dept of Medical Sciencies, Uppsala University, Uppsala, Sweden
Locations (6):
- Sweden (6):
  - Gastroenterology department, Falun
  - Gastroenterology outpatientclinic, Sahlgrenska hospital, Gothenburg
  - Gastroenterology outpatient department, Skane Universityhospital, Malmo
  - Gastroenterology department, Örebro Universityhospital, Örebro
  - Gastroenterology department, Danderyd hospital, Stockholm
  - Gastroenterology department, Uppsala academical hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from Region Dalarna upon reasonable request, provided that the data can be made available in accordance with applicable data protection and privacy regulations.
  Contact information: Maria Hjorth, maria.hjorth@regiondalarna.se and diariet@regiondalarna.se

REFERENCES:
- [Background] Arguedas MR, DeLawrence TG, McGuire BM. Influence of hepatic encephalopathy on health-related quality of life in patients with cirrhosis. Dig Dis Sci. 2003 Aug;48(8):1622-6. doi: 10.1023/a:1024784327783. PMID 12924658
- [Background] Abdi F, Daryani NE, Khorvash F, Yousefi Z. Experiences of Individuals With Liver Cirrhosis: A Qualitative Study. Gastroenterol Nurs. 2015 Jul-Aug;38(4):252-7. doi: 10.1097/SGA.0000000000000122. PMID 26226019
- [Background] Arvidsson SB, Petersson A, Nilsson I, Andersson B, Arvidsson BI, Petersson IF, Fridlund B. A nurse-led rheumatology clinic's impact on empowering patients with rheumatoid arthritis: A qualitative study. Nurs Health Sci. 2006 Sep;8(3):133-9. doi: 10.1111/j.1442-2018.2006.00269.x. PMID 16911172
- [Background] Biddle ML, Adler NR, Heath M, Streat S, Wardrop M, Watson JP. Nurse-led clinic: effective and efficient delivery of assessment and review of patients with hepatitis B and C. Intern Med J. 2014 Jun;44(6):581-5. doi: 10.1111/imj.12400. PMID 24612294
- [Background] Bleibel W, Al-Osaimi AM. Hepatic encephalopathy. Saudi J Gastroenterol. 2012 Sep-Oct;18(5):301-9. doi: 10.4103/1319-3767.101123. PMID 23006457
- [Background] Borhofen SM, Gerner C, Lehmann J, Fimmers R, Gortzen J, Hey B, Geiser F, Strassburg CP, Trebicka J. The Royal Free Hospital-Nutritional Prioritizing Tool Is an Independent Predictor of Deterioration of Liver Function and Survival in Cirrhosis. Dig Dis Sci. 2016 Jun;61(6):1735-43. doi: 10.1007/s10620-015-4015-z. Epub 2016 Jan 2. PMID 26725059
- [Background] Brown MT, Bussell JK. Medication adherence: WHO cares? Mayo Clin Proc. 2011 Apr;86(4):304-14. doi: 10.4065/mcp.2010.0575. Epub 2011 Mar 9. PMID 21389250
- [Background] Chaney A, Werner KT & Kipple T. Primary care management of hepatic encephalopathy: A common cirrhosis complication. The journal for Nurse Practisioners. 11(3): 300-306, 2015.
- [Background] Disler RT, Gallagher RD, Davidson PM. Factors influencing self-management in chronic obstructive pulmonary disease: an integrative review. Int J Nurs Stud. 2012 Feb;49(2):230-42. doi: 10.1016/j.ijnurstu.2011.11.005. Epub 2011 Dec 6. PMID 22154095
- [Background] Evangelista LS, Shinnick MA. What do we know about adherence and self-care? J Cardiovasc Nurs. 2008 May-Jun;23(3):250-7. doi: 10.1097/01.JCN.0000317428.98844.4d. PMID 18437067
- [Background] Hays RD, Morales LS. The RAND-36 measure of health-related quality of life. Ann Med. 2001 Jul;33(5):350-7. doi: 10.3109/07853890109002089. PMID 11491194
- [Background] Hommel A, Idvall E & Andersson AC. Kvalitetsutveckling: Kvalitet och omvårdnad. I AK Edberg, A Ehrenberg, F Friberg, L Wallin, H Wijk & J Öhlén (Eds) Omvårdnad på avancerad nivå: Kärnkompetenser inom sjuksköterskans specialistområden (1st ed, pp. 147-150), 2013.
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Infante-Rivard C, Esnaola S, Villeneuve JP. Clinical and statistical validity of conventional prognostic factors in predicting short-term survival among cirrhotics. Hepatology. 1987 Jul-Aug;7(4):660-4. doi: 10.1002/hep.1840070408. PMID 3610046
- [Background] Jahren Kristoffersen N, Nortveldt F & Skaug EA. Grundläggande omvårdnad del 1. Stockholm: Liber AB, 2005.
- [Background] Jones JC, Coombes JS, Macdonald GA. Exercise capacity and muscle strength in patients with cirrhosis. Liver Transpl. 2012 Feb;18(2):146-51. doi: 10.1002/lt.22472. PMID 22139897
- [Background] Jorgensen R. A phenomenological study of fatigue in patients with primary biliary cirrhosis. J Adv Nurs. 2006 Sep;55(6):689-97. doi: 10.1111/j.1365-2648.2006.03958.x. PMID 16925617
- [Background] Kalaitzakis E, Josefsson A, Bjornsson E. Type and etiology of liver cirrhosis are not related to the presence of hepatic encephalopathy or health-related quality of life: a cross-sectional study. BMC Gastroenterol. 2008 Oct 15;8:46. doi: 10.1186/1471-230X-8-46. PMID 18922174
- [Background] Kamath PS, Wiesner RH, Malinchoc M, Kremers W, Therneau TM, Kosberg CL, D'Amico G, Dickson ER, Kim WR. A model to predict survival in patients with end-stage liver disease. Hepatology. 2001 Feb;33(2):464-70. doi: 10.1053/jhep.2001.22172. PMID 11172350
- [Background] Kirkevold M. Omvårdnadsteorier; Analys och utvärdering (2nd Ed). Lund: Studentlitteratur, 2000.
- [Background] Koay K, Schofield P, Jefford M. Importance of health literacy in oncology. Asia Pac J Clin Oncol. 2012 Mar;8(1):14-23. doi: 10.1111/j.1743-7563.2012.01522.x. PMID 22369440
- [Background] Kroese ME, Severens JL, Schulpen GJ, Bessems MC, Nijhuis FJ, Landewe RB. Specialized rheumatology nurse substitutes for rheumatologists in the diagnostic process of fibromyalgia: a cost-consequence analysis and a randomized controlled trial. J Rheumatol. 2011 Jul;38(7):1413-22. doi: 10.3899/jrheum.100753. Epub 2011 Apr 1. PMID 21459951
- [Background] Larsson, B, Larsson G, Larsson M & Starrin B. KUPP-boken: Vägledning till frågeformuläret KUPP, Kvalitet ur patientperspektiv. Stockholm: Grafiska Gruppen, 2001.
- [Background] Larsson G, Larsson BW, Munck IM. Refinement of the questionnaire 'quality of care from the patient's perspective' using structural equation modelling. Scand J Caring Sci. 1998;12(2):111-8. PMID 9801632
- [Background] Maldonado-Garza HJ, Vazquez-Elizondo G, Gaytan-Torres JO, Flores-Rendon AR, Cardenas-Sandoval MG, Bosques-Padilla FJ. Prevalence of minimal hepatic encephalopathy in cirrhotic patients. Ann Hepatol. 2011 Jun;10 Suppl 2:S40-4. PMID 22228880
- [Background] Nardelli S, Pentassuglio I, Pasquale C, Ridola L, Moscucci F, Merli M, Mina C, Marianetti M, Fratino M, Izzo C, Merkel C, Riggio O. Depression, anxiety and alexithymia symptoms are major determinants of health related quality of life (HRQoL) in cirrhotic patients. Metab Brain Dis. 2013 Jun;28(2):239-43. doi: 10.1007/s11011-012-9364-0. Epub 2013 Jan 8. PMID 23296469
- [Background] Pasqualetti P, Di Lauro G, Festuccia V, Giandomenico G, Casale R. Prognostic value of Pugh's modification of Child-Turcotte classification in patients with cirrhosis of the liver. Panminerva Med. 1992 Apr-Jun;34(2):65-8. PMID 1408330
- [Background] Prytz H & Ståhl P. Levercirros och dess kliniska manifestationer. I R Hultcrantz, A Bergquist, S Lindgren, M Simrén, P Stål & OB Suhr (Eds.). Gastroenterologi och hepatologi. Stockholm: Liber. (1st ed, pp. 451-475), 2011.
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Riley TR, Taheri M, Schreibman IR. Does weight history affect fibrosis in the setting of chronic liver disease? J Gastrointestin Liver Dis. 2009 Sep;18(3):299-302. PMID 19795023
- [Background] Schadewaldt V, Schultz T. Nurse-led clinics as an effective service for cardiac patients: results from a systematic review. Int J Evid Based Healthc. 2011 Sep;9(3):199-214. doi: 10.1111/j.1744-1609.2011.00217.x. PMID 21884449
- [Background] Shen C, Zhao CY, Zhang R, Qiao L. Obesity-related hepatocellular carcinoma: roles of risk factors altered in obesity. Front Biosci (Landmark Ed). 2012 Jun 1;17(6):2356-70. doi: 10.2741/4057. PMID 22652784
- [Background] Sheridan SL, Halpern DJ, Viera AJ, Berkman ND, Donahue KE, Crotty K. Interventions for individuals with low health literacy: a systematic review. J Health Commun. 2011;16 Suppl 3:30-54. doi: 10.1080/10810730.2011.604391. PMID 21951242
- [Background] Shutt JD, Robathan J, Vyas SK. Impact of a clinical nurse specialist on the treatment of chronic hepatitis C. Br J Nurs. 2008 May 8-21;17(9):572-5. doi: 10.12968/bjon.2008.17.9.29242. PMID 18562991
- [Background] Volk ML, Fisher N, Fontana RJ. Patient knowledge about disease self-management in cirrhosis. Am J Gastroenterol. 2013 Mar;108(3):302-5. doi: 10.1038/ajg.2012.214. PMID 23459041
- [Background] Wakim-Fleming J, Mullen KD. Long-term management of alcoholic liver disease. Clin Liver Dis. 2005 Feb;9(1):135-49. doi: 10.1016/j.cld.2004.10.001. PMID 15763233
- [Background] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308
- [Background] Wiesner R, Edwards E, Freeman R, Harper A, Kim R, Kamath P, Kremers W, Lake J, Howard T, Merion RM, Wolfe RA, Krom R; United Network for Organ Sharing Liver Disease Severity Score Committee. Model for end-stage liver disease (MELD) and allocation of donor livers. Gastroenterology. 2003 Jan;124(1):91-6. doi: 10.1053/gast.2003.50016. PMID 12512033
- [Background] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Background] Weissenborn K, Ennen JC, Schomerus H, Ruckert N, Hecker H. Neuropsychological characterization of hepatic encephalopathy. J Hepatol. 2001 May;34(5):768-73. doi: 10.1016/s0168-8278(01)00026-5. No abstract available. PMID 11434627
- [Background] Wigg AJ, McCormick R, Wundke R, Woodman RJ. Efficacy of a chronic disease management model for patients with chronic liver failure. Clin Gastroenterol Hepatol. 2013 Jul;11(7):850-8.e1-4. doi: 10.1016/j.cgh.2013.01.014. Epub 2013 Jan 29. PMID 23375997
- [Background] Wilde B, Starrin B, Larsson G, Larsson M. Quality of care from a patient perspective--a grounded theory study. Scand J Caring Sci. 1993;7(2):113-20. doi: 10.1111/j.1471-6712.1993.tb00180.x. PMID 8248668
- [Background] Wilde Larsson B, Larsson G. Development of a short form of the Quality from the Patient's Perspective (QPP) questionnaire. J Clin Nurs. 2002 Sep;11(5):681-7. doi: 10.1046/j.1365-2702.2002.00640.x. PMID 12201896
- [Derived] Hjorth M, Sjoberg D, Svanberg A, Lo Martire R, Kaminsky E, Rorsman F. Health-related quality of life in patients with liver cirrhosis following adjunctive nurse-based care versus standard medical care: a pragmatic, multicentre, randomised controlled study. BMJ Open Gastroenterol. 2025 Jan 31;12(1):e001694. doi: 10.1136/bmjgast-2024-001694. PMID 39890127
- [Derived] Hjorth M, Svanberg A, LoMartire R, Kaminsky E, Rorsman F. Patient perceived quality of cirrhosis care- adjunctive nurse-based care versus standard medical care: a pragmatic multicentre randomised controlled study. BMC Nurs. 2024 Apr 19;23(1):251. doi: 10.1186/s12912-024-01934-9. PMID 38637755
- [Derived] Hjorth M, Sjoberg D, Svanberg A, Kaminsky E, Langenskiold S, Rorsman F. Nurse-led clinic for patients with liver cirrhosis-effects on health-related quality of life: study protocol of a pragmatic multicentre randomised controlled trial. BMJ Open. 2018 Oct 17;8(10):e023064. doi: 10.1136/bmjopen-2018-023064. PMID 30337316
- See also: Practice Guideline by the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases. (2014). Hepatic encephalopathy in chronic liver disease. — http://www.easl.eu/medias/cpg/Hepatic-Encephalopathy-Chronic-Liver-Disease/English-report.pdf
- See also: Swedish Code of Statutes 1982:763. Swedish health care act. Retrieved from the Swedish parliament — http://www.riksdagen.se/sv/Dokument-Lagar/Lagar/Svenskforfattningssamling/Halso--och-sjukvardslag-1982_sfs-1982-763/
- See also: Swedish Code of Statutes 1998:204. Swedish Personal Data Act. Retrieved from the Swedish parliament — http://www.riksdagen.se/sv/Dokument-Lagar/Lagar/Svenskforfattningssamling/Personuppgiftslag-1998204_sfs-1998-204/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT02957253/Prot_SAP_ICF_000.pdf